CLINICAL TRIAL: NCT05707338
Title: Short-term Outcomes of Laparoscopic Versus Open Gastrectomy With Lymph Node Dissection for Early Gastric Cancer :a Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Nasser Mohamed Ali, assisstant lecturer of general surgery department, Sohag university hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-01-16
Record Dates: First submitted 2023-01-22; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Early Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy; Lymph Node Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic group (Active Comparator)
  Interventions: Procedure: Gastrectomy with lymph node dissection
- open group (Active Comparator)
  Interventions: Procedure: Gastrectomy with lymph node dissection

INTERVENTIONS:
Procedure: Gastrectomy with lymph node dissection — prospective randomized comparative clinical trial study analyzing outcomes of gastrectomy for early gastric cancer using laporoscopy versus open approach. This will be a prospective comparative study at Sohag University Hospital, Egypt and National Cancer Institute(NCI), Cairo university ,Egypt.
  Patients were divided randomizly into two groups; the first group included patients who will have laparoscopic gastrectomy (Lap group), and the second group included patients will receive open gastrectomy (Open group).

SUMMARY:
While the incidence of gastric cancer is gradually declining, it is the fifth most common cancer worldwide and the third most common cause of cancer related death worldwide according to GLOBOCAN 2018 data (Rawla P and Barsouk A.,2019).

Laparoscopic distal gastrectomy for early gastric cancer(EGC) was first performed more than 20 years ago (Shi, Y et al.,2018). Laparoscopy-assisted gastrectomy (LAG) for EGC has been confirmed to have oncologic and long-term survival equivalency to the open technique and provide tremendous advantages over open surgery, such as good cosmesis, reduced pain, and shorter hospital stay(Katai H et al.,2017).

Based on the experience of EGC, most experienced surgeons have applied the laparoscopic procedure in patients with locally advanced gastric cancer (AGC). Retrospective studies have assessed the technical and oncological safety of LAG with D2 lymph node dissection for AGC(Hao Y et al .,2016).

Recently, results of two ongoing randomized controlled trials (RCTs) have revealed the surgical safety of laparoscopic distal gastrectomy with D2 lymphadenectomy for AGC . However, laparoscopic gastrectomy for locally advanced disease remains controversial(Hu Y et al.,2016).

Here, we report the short-term surgical outcomes of a RCT comparing laparoscopic and open gastrectomy (OG) with D2 lymph node dissection for EGC, which was designed to assess the technical safety and oncologic feasibility of LAG for EGC.

DETAILED DESCRIPTION:
Aim of the work

a prospective randomized controlled trial comparing laparoscopic and open gastrectomy with D2 lymph node dissection for EGC to evaluate technical safety and oncologic feasibility.

The postoperative morbidity and mortality rates will be based on the modified intention-to-treat analysis.

The aim of this study is to compare the operative and short-term oncologic outcomes of laparoscopic versus open resections.

Patients and methods

The study design: : prospective randomized comparative clinical trial study analyzing outcomes of gastrectomy for early gastric cancer using laporoscopy versus open approach. This will be a prospective comparative study at Sohag University Hospital, Egypt and National Cancer Institute(NCI), Cairo university ,Egypt.

Patients were divided randomizly into two groups; the first group included patients who will have laparoscopic gastrectomy (Lap group), and the second group included patients will receive open gastrectomy (Open group).

Study population

The study included patients complaining of gastric cancer stage (T1-T2N0M0).The study will start from december 2022 .

Inclusion criteria: Inclusion criteria were as follows: histologically confirmed adenocarcinoma of the stomach; pathologically confirmed stage T1-T2; no evidence of distant metastasis by means of abdominal computed tomography(CECT) and CT chest ; D2 lymphadenectomy with curative R0

according to pathological diagnosis after the operation . patients with N1 confirmed pathologically after operation also will be included in the study.

The exclusion criteria:

1. pregnancy
2. an American Society of Anesthesiologists (ASA) score > 3,
3. severe mental disorders
4. prior upper abdominal surgery except laparoscopic cholecystectomy,
5. presence of other malignancies
6. a history of chemotherapy or radiation therapy.
7. unstable angina or myocardial infarction within the past 6 months, severe respiratory disease (forced expiratory volume in 1 s, FEV1 < 50%)
8. abdominal wall hernia
9. diaphragmatic hernia
10. coagulation disorder
11. portal hypertension
12. Advanced gastric cancer (stage;T3,T4,N1 to 3 ,M1) based on preoperative diagnosis.

Approvals and consents

This study will be done after obtaining approval from the research ethics committee of the Sohag faculty of medicine. A written Informed consent will be obtained from all participants before being enrolled in the study and before performing the procedure after receiving an explanation of the study protocol, including both types of operation and possible complications. The study will be registered at www.clinicaltrials.gov.

Data collection:

Registered data will be collected from the hospital databases, clinical data.

Randomization

Randomization was performed by closed envelopes and was balanced and stratified for proposed type of resection.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients complaining of gastric cancer stage (T1-T2N0M0).The study will start from december 2022 .

Inclusion criteria: Inclusion criteria were as follows: histologically confirmed adenocarcinoma of the stomach; pathologically confirmed stage T1-T2; no evidence of distant metastasis by means of abdominal computed tomography(CECT) and CT chest ; D2 lymphadenectomy with curative R0

according to pathological diagnosis after the operation . patients with N1 confirmed pathologically after operation also will be included in the study.

Exclusion Criteria:

1. pregnancy
2. an American Society of Anesthesiologists (ASA) score > 3,
3. severe mental disorders
4. prior upper abdominal surgery except laparoscopic cholecystectomy,
5. presence of other malignancies
6. a history of chemotherapy or radiation therapy.
7. unstable angina or myocardial infarction within the past 6 months, severe respiratory disease (forced expiratory volume in 1 s, FEV1 < 50%)
8. abdominal wall hernia
9. diaphragmatic hernia
10. coagulation disorder
11. portal hypertension
12. Advanced gastric cancer (stage;T3,T4,N1 to 3 ,M1) based on preoperative diagnosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
early postoperative complications | 20 month

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hao Y, Yu P, Qian F, Zhao Y, Shi Y, Tang B, Zeng D, Zhang C. Comparison of laparoscopy-assisted and open radical gastrectomy for advanced gastric cancer: A retrospective study in a single minimally invasive surgery center. Medicine (Baltimore). 2016 Jun;95(25):e3936. doi: 10.1097/MD.0000000000003936. PMID 27336885
- [Background] Hu Y, Huang C, Sun Y, Su X, Cao H, Hu J, Xue Y, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Chen P, Liu H, Zheng C, Liu F, Yu J, Li Z, Zhao G, Chen X, Wang K, Li P, Xing J, Li G. Morbidity and Mortality of Laparoscopic Versus Open D2 Distal Gastrectomy for Advanced Gastric Cancer: A Randomized Controlled Trial. J Clin Oncol. 2016 Apr 20;34(12):1350-7. doi: 10.1200/JCO.2015.63.7215. Epub 2016 Feb 22. PMID 26903580
- [Background] Katai H, Mizusawa J, Katayama H, Takagi M, Yoshikawa T, Fukagawa T, Terashima M, Misawa K, Teshima S, Koeda K, Nunobe S, Fukushima N, Yasuda T, Asao Y, Fujiwara Y, Sasako M. Short-term surgical outcomes from a phase III study of laparoscopy-assisted versus open distal gastrectomy with nodal dissection for clinical stage IA/IB gastric cancer: Japan Clinical Oncology Group Study JCOG0912. Gastric Cancer. 2017 Jul;20(4):699-708. doi: 10.1007/s10120-016-0646-9. Epub 2016 Oct 7. PMID 27718137
- [Background] Shi Y, Xu X, Zhao Y, Qian F, Tang B, Hao Y, Luo H, Chen J, Yu P. Short-term surgical outcomes of a randomized controlled trial comparing laparoscopic versus open gastrectomy with D2 lymph node dissection for advanced gastric cancer. Surg Endosc. 2018 May;32(5):2427-2433. doi: 10.1007/s00464-017-5942-x. Epub 2017 Dec 12. PMID 29234941